CLINICAL TRIAL: NCT02818478
Title: Patient Reported Outcome Measures Reported Into the Danish Arthritis Registry (DANBIO) Via Computer or Tablet at Home Versus Touch Screen at the Outpatient Clinic Among Patients With Axial Spondyloarthritis or Rheumatoid Arthritis
Brief Title: Patient Reported Outcomes Reported Via PC / Tablet Home Versus Touch Screen at Hospital Among Patients With Arthritis
Acronym: PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henrik Gudbergsen (Other)
Collaborators: The DANBIO registry, Denmark (Unknown); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Henrik Gudbergsen, EU Project Coordinator, Parker Research Institute
Organization: Parker Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 100.03
Record Dates: First submitted 2016-05-23; First posted 2016-06-29 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis; Axial Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RA; at home first (Other): Patients in this arm (10 patients with rheumatoid arthirtis, RA) will be randomised to initially fill in patient reported outcome measures from home via their own computer or tablet; subsequently these patients will fill in patient reported outcome measures at the outpatient clinic
  Interventions: Other: Reporting of patient reported outcome measures
- RA; outpatient clinic first (Other): Patients in this arm (10 patients with rheumatoid arthirtis, RA) will be randomised to initially fill in patient reported outcome measures at the outpatient clinic; subsequently these patients will fill in patient reported outcome measures from home via their own computer or tablet
  Interventions: Other: Reporting of patient reported outcome measures
- AxSpa; at home first (Other): Patients in this arm (10 patients with axial spondyloarthritis, AxSpa) will be randomised to initially fill in patient reported outcome measures from home via their own computer or tablet; subsequently these patients will fill in patient reported outcome measures at the outpatient clinic
  Interventions: Other: Reporting of patient reported outcome measures
- AxSpa; outpatient clinic first (Other): Patients in this arm (10 patients with axial spondyloarthritis, AxSpa) will be randomised to initially fill in patient reported outcome measures at the outpatient clinic; subsequently these patients will fill in patient reported outcome measures from home via their own computer or tablet
  Interventions: Other: Reporting of patient reported outcome measures

INTERVENTIONS:
Other: Reporting of patient reported outcome measures — Electronic reporting of patient reported outcome measures from home, compared to reporting of patient reported outcome measures at the outpatient clinic

SUMMARY:
To investigate if electronic reporting of patient reported outcome measures from home is comparable to the traditional touch-screen solution to hospital among patients with rheumatoid arthritis and axial spondyloarthritis

ELIGIBILITY:
Inclusion Criteria

* Rheumatoid arthirtis OR axial spondyloarthritis
* Active treatment and monitoring of the Knowledge Center for Rheumatology and Spine diseases, Rigshospitalet, Denmark
* Patients must have reported patient reported outcome measures via DANBIOs touch-screen solution ≥ 3 times

Exclusion Criteria

* Impaired vision
* Non-Danish speaking
* No electronic device at home,, tablet or computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HAQ | 48 hours
  The Health Assessment Questionnaire (HAQ) developed to retrieve quantitative information on outcomes among patients with rheumatoid arthritis

SECONDARY OUTCOMES:
100 mm VAS global | 48 hours
  Assessed via a visual analogue scale (VAS)
100 mm VAS pain | 48 hours
  Assessed via a visual analogue scale (VAS)
100 mm VAS fatigue | 48 hours
  Assessed via a visual analogue scale (VAS)
BASDAI | 48 hours
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) developed to retrieve quantitative information on outcomes among patients with Ankylosing Spondylitis
BASFI | 48 hours
  The Bath Ankylosing Spondylitis Functional Index (BASFI) developed to retrieve quantitative information on outcomes among patients with Ankylosing Spondylitis
BASDAI 5 & 6 | 48 hours
  Questions 5 and 6 in BASDAI

OTHER OUTCOMES:
Smoking questionnaire | 48 hours
  Smoking habits (I currently smoke; if smoking, then how many cigarettes, pibes, cigarillos, cigars and/or cheroots per day / I smoke from time to time; less than 1 cigarettes, or an equivalent amount, per day / I have stopped smoking; year of cessation / I have never smoked)
Alcohol consumption (units consumed per week) | 48 hours
Exercise questionnaire | 48 hours
  Level of exercise; "exercise that causes an increased pulse and/or a feeling of being breathless" (5 times per week / 3-4 times per week / 1-2 times per week / 1-2 times per month / no regular exercising / I do not exercise)
Medical conditions questionnaire | 48 hours
  Diagnosis of other medical conditions; "Has a doctor ever said that you have or have had the following diseases?" (hypertension / diabetes / tuberculosis / angina / hypercholesterolemia / heart attack / brain haemorrhage / asthma / psoriasis / chronic bronchitis / osteoporosis / ulcer / liver disease / kidney disease / depression / inflammatory bowel disease or Crohns disease / cancer / multiple sclerosis / thyroid disease)

CONTACTS AND LOCATIONS:
Overall Officials: Merete M Hetland, MD.PhD.DMSc, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No